CLINICAL TRIAL: NCT05427162
Title: Open-Label, Randomized Study to Evaluate Safety, Tolerability, and Pharmacokinetics of Single and Multiple Doses of Different Formulations of an IP Receptor Agonist
Brief Title: A Study of Single and Multiple Doses of Different Formulations of a Prostacyclin Receptor Agonist
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Actelion (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CR109201
Record Dates: First submitted 2022-06-16; First posted 2022-06-22 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Pulmonary Arterial Hypertension
MeSH Terms: conditions — Pulmonary Arterial Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Prostacyclin Receptor Agonist (Experimental): Participants in Cohort 1-7 will receive multiple doses of prostacyclin receptor agonist of formulation 1 in treatment period 1, followed by a single dose of various other formulations (formulation 2, 3, and 4) in treatment period 2. Cohort 7 will be optional. Doses in Cohorts 4, 5, 6 and cohort 7 will be based on PK, safety and tolerability data of previous 3 cohorts (preceding cohorts).
  Interventions: Drug: Prostacyclin Receptor Agonist

INTERVENTIONS:
Drug: Prostacyclin Receptor Agonist — Prostacyclin receptor agonist will be administered.

SUMMARY:
The purpose of the study is to assess safety and tolerability of prostacyclin receptor agonist formulation in treatment period 1 and with different formulation of prostacyclin receptor agonist in treatment period 2.

ELIGIBILITY:
Inclusion Criteria:

* Otherwise, healthy as deemed by the investigator on the basis of physical examination, medical history, vital signs, and 12-lead electrocardiograms (ECG) performed at Screening and Day -1 of oral treatment period
* Otherwise, healthy medically stable on the basis of clinical laboratory tests performed at screening. If the results of the serum chemistry panel, blood coagulation, hematology, or urinalysis are outside the normal reference ranges, the participant may be included only if the investigator judges the abnormalities or deviations from normal to be not clinically significant or to be appropriate and reasonable for the population under study. This determination must be recorded in the participant's source documents and initialed by the investigator
* Body mass index (BMI) within the range 18.0 to 32.0 kilograms per meter square (kg/m^2) (inclusive) and body weight not less than 50 kilograms (kg) at screening
* All female participants must have a negative highly sensitive serum (beta-human chorionic gonadotropin [beta-hCG]) at screening
* A male participant must agree not to donate sperm for the purpose of reproduction during the study and for a minimum of 90 days after receiving the last dose of study intervention

Exclusion Criteria:

* Known allergies, hypersensitivity, anaphylaxis, or intolerance to prostacyclin receptor agonist or drugs of the same class, or any excipient (including poloxamer and polysorbate) of the drug formulation(s)
* Clinically significant abnormal physical examination, vital signs, or 12-lead ECG (QTc greater than or equal to [>=]450 milliseconds [msec] for men and >=460 msec for women. QT corrected according to Bazett's formula [QTcB]) as assessed by the Investigator at Screening or Day -1 of oral treatment period
* History of malignancy within 3 years before screening (exceptions are squamous and basal cell carcinomas of the skin
* Positive serologic testing for human immunodeficiency virus (HIV), hepatitis B surface antigen (hBsAg), hepatitis C virus (HCV), active coronavirus disease 2019 (COVID-19) infection
* A history of repeated (more than once over the last 30 days) fainting due to cardiac cause, collapse, syncope, orthostatic hypotension, or vasovagal reactions

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 88 (Actual)
Dates: Start 2022-06-21 (Actual); Primary Completion 2023-12-05 (Actual); Study Completion 2023-12-05 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Treatment-emergent Adverse Events (TEAEs) | Up to 114 days
  An adverse event is any untoward medical event that occurs in a participant administered an investigational product, and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product. TEAEs are defined as AEs with onset or worsening on or after date of first dose of study treatment.
Number of Participants With Serious TEAEs | Up to 114 days
  A SAE is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Serious TEAEs are defined as serious events between administration of study drug and after the last dose that were absent before treatment or that worsen relative to pretreatment state.
Number of Participants with TEAEs by Severity | Up to 114 days
  Number of participants with TEAEs by severity will be evaluated. An assessment of severity grade will be made using the following general categorical descriptors, such as Mild (Awareness of symptoms that are easily tolerated, causing minimal discomfort, and not interfering with everyday activities), Moderate (Sufficient discomfort is present to cause interference with normal activity), and Severe (Extreme distress, causing significant impairment of functioning or incapacitation, and prevents normal everyday activities).
Number of Participants with TEAEs Leading to Discontinuation | Up to 114 days
  Number of participants with TEAEs leading to discontinuation will be reported.
Number of Participants With Change from Baseline in Clinical Laboratory Values | Up to 114 days
  Number of participants with change from baseline in clinical laboratory values (chemistry, hematology, and urinalysis) will be evaluated.
Number of Participants With Injection Site Reactions | Up to 114 days
  Number of participants with injection site reactions will be evaluated.

SECONDARY OUTCOMES:
Treatment Period 1: Maximum Observed Plasma Concentration of Prostacyclin Receptor Agonist at Steady State (Cmax[ss]) | Up to 114 days
  Cmax(ss) is the maximum observed plasma concentration of prostacyclin receptor agonist at steady state, during treatment period 1.
Treatment Period 1: Time to Reach Maximum Observed Plasma Concentration of Prostacyclin Receptor Agonist at Steady State (Tmax[ss]) | Up to 114 days
  Tmax(ss) is the actual sampling time to reach maximum observed plasma concentration of prostacyclin receptor agonist at steady state, during treatment period 1.
Treatment Period 1: Area Under the Curve From Time Zero to tau of Prostacyclin Receptor Agonist at Steady State (AUC[0-tau{ss}]) | Up to 114 days
  AUC(0-tau[ss]) is defined as area under the curve from time 0 to tau hours post dose of prostacyclin receptor agonist at steady state, during treatment period 1.
Treatment Period 1: Plasma Concentration at the End of One Dose Interval of Prostacyclin Receptor Agonist at Steady State (Ctrough[ss]) | Up to 114 days
  Ctrough(ss) is the plasma concentration at the end of one dose interval of prostacyclin receptor agonist at steady state, during treatment period 1.
Treatment Period 2: Maximum Observed Plasma Concentration (Cmax) of Prostacyclin Receptor Agonist | Up to 114 days
  Cmax is the maximum observed plasma concentration of prostacyclin receptor agonist, during treatment period 2.
Treatment Period 2: Time to Reach Maximum Observed Plasma Concentration (Tmax) of Prostacyclin Receptor Agonist | Up to 114 days
  Tmax is the actual sampling time to reach maximum observed plasma concentration of prostacyclin receptor agonist, during treatment period 2.
Treatment Period 2: Area Under the Plasma Concentration-time Curve from time Zero to time t (AUC[0-t]) of Prostacyclin Receptor Agonist | Up to 114 days
  Area under the plasma concentration-time curve from time zero to time t of the last measured concentration above the limit of concentration of prostacyclin receptor agonist, during treatment period 2.
Treatment Period 2: Area Under the Plasma Concentration Time Curve From Time Zero to Infinite Time (AUC [0-infinity]) of Prostacyclin Receptor Agonist | Up to 114 days
  AUC (0-infinity) is the area under the plasma concentration-time curve from time zero to infinite time calculated as the sum of AUC (0-last) and C (0-last)/ lambda(z); wherein AUC (0-last) is area under the plasma concentration time curve from time zero to last quantifiable time, C(0-last) is the last observed quantifiable concentration of prostacyclin receptor agonist, and lambda (z) is elimination rate constant, during treatment period 2.
Treatment Period 2: Area Under the Plasma Concentration-time Curve From Zero to Time 24 Hours (AUC [0-24h]) of Prostacyclin Receptor Agonist | Predose up to 24 hours post dose
  AUC (0-24h) is the area under the plasma concentration-time curve from zero to time 24 hours, during treatment period 2.
Treatment Period 2: Area Under the Plasma Concentration-time Curve From Zero to Day 14 (AUC [0-Day 14]) of Prostacyclin Receptor Agonist | Up to Day 14
  AUC (0-Day 14) is the area under the plasma concentration-time curve from zero to Day 14, during treatment period 2.
Treatment Period 2: Area Under the Plasma Concentration-time Curve From Zero to Day 28 (AUC [0-Day 28]) of Prostacyclin Receptor Agonist | Up to Day 28
  AUC (0-Day 28) is the area under the plasma concentration-time curve from zero to Day 28, during treatment period 2.
Treatment Period 2: Plasma Concentration of Prostacyclin Receptor Agonist at Day 14 (C[Day 14]) | Up to Day 14
  C(Day 14) is the plasma concentration of prostacyclin receptor agonist at Day 14, during treatment period 2
Treatment Period 2: Plasma Concentration of Prostacyclin Receptor Agonist at Day 28 (C[Day 28]) | Up to Day 28
  C(Day 28) is the plasma concentration of prostacyclin receptor agonist at Day 28, during treatment period 2.

CONTACTS AND LOCATIONS:
Overall Officials: Actelion Pharmaceuticals Ltd. Clinical Trials, Study Director — Actelion
Locations (1):
- Celerion, Tempe, Arizona, United States

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: http://www.janssen.com/clinical-trials/transparency